CLINICAL TRIAL: NCT00626782
Title: Lucentis Versus Mitomycin C as Adjunctive Agent During Trabeculectomy Surgery
Brief Title: Lucentis Versus Mitomycin C During Glaucoma Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Genentech, Inc. (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Michael Pro, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#07-819; rhuFAB v2 (Other Grant/Funding Number: Genentec)
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Glaucoma
Keywords: glaucoma; glucoma filtering surgery; ranibizumab; mitomycin C; patients requiring first time glaucoma filtering surgery
MeSH Terms: conditions — Glaucoma | interventions — Ranibizumab; Mitomycin

STUDY DESIGN:
Intervention Model Description: Patients requiring trabeculectomy were randomly assigned to either MMC or Ranibizumab during surgery.
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Ranibizumab 0.5mg (0.05mL) injection (Experimental): Ranibizumab 0.5mg (0.05mL) injection at end of trabeculectomy surgery. This intra-operative adjunct therapy was administered sub-conjunctivally 8-10mm posteriorly to the limbus as an antifibrotic agent.
  Interventions: Drug: Ranibizumab
- B: Mitomycin C 0.4 mg/ml sponge (Active Comparator): Mitomycin C 0.4 mg/ml soaked sponge applied to sclera (for up to 2 min) after flap is made during trabeculectomy surgery. This is the typical method used as an antifibrotic agent.
  Interventions: Drug: Mitomycin (MMC)

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab 0.5mg (0.05mL)one injection in sub-tenon's at the conclusion of glaucoma surgery
  Other Names: Lucentis
  Arms: A: Ranibizumab 0.5mg (0.05mL) injection
Drug: Mitomycin (MMC) — Mitomycin (MMC) C 0.4 mg/ml applied with soaked pledget inserted in the sub-tenon's space during glaucoma surgery.
  Other Names: MMC C 0.4 mg/ml
  Arms: B: Mitomycin C 0.4 mg/ml sponge

SUMMARY:
Does a new add on (or adjunctive) therapy used in glaucoma surgery improve the success of trabeculectomy? Ranibizumab may offer benefit similar to mitomycin C in preventing epi-scleral fibrosis while avoiding the well known complications of mytomycin C which include late bleb leaks, hypotony and infection.

DETAILED DESCRIPTION:
This is an open-label, single center trial with two arms for patients who underwent guarded filtration surgery to control glaucoma. The control will consist of patients randomly assigned to receive inter-operative mitomycin C 0.4 mg/ml which is applied in a standard fashion with a soaked pledget inserted in the sub-tenon's space during surgery. The study arm will consist of patients randomly assigned to receive a sub-tenon injection of Ranibizumab 0.5 mg/0.05mL with a 30 gauge needle on a tuberculin syringe at the termination of the surgery. No mitomycin C will be applied.

Post operative follow-up will consist of a minimum of 6 visits during a one year period.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs or older
* patients requiring first time glaucoma filtering surgery
* phakic or pseudophakic
* must provide written informed consent and comply with study assignments

Exclusion Criteria:

* Pregnant, lactation or premenopausal women not using adequate contraception.
* Previous glaucoma surgery, tube shunt surgery, pars plana vitrectomy, scleral buckle, penetrating keratoplasty.
* Abnormality preventing reliable applanation tonometry in each eye.
* Current infection or inflammation in either eye.
* Enrolled in another investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Pro, MD, Principal Investigator — Wills Eye Institute
Locations (1):
- Wills Eye Hospital, Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pro MJ, Freidl KB, Neylan CJ, Sawchyn AK, Wizov SS, Moster MR. Ranibizumab versus mitomycin C in primary trabeculectomy--a pilot study. Curr Eye Res. 2015 May;40(5):510-5. doi: 10.3109/02713683.2014.935441. Epub 2014 Jul 14. PMID 25019269

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment 1 (Ranibizumab 0.5mg): Ranibizumab 0.5mg (0.05mL) injection at end of trabeculectomy surgery.
  Ranibizumab: Ranibizumab 0.5mg (0.05mL)one injection in sub-tenon's at the conclusion of glaucoma surgery
- Treatment 2 (Mitomycin C 0.4 mg/ml): Mitomycin C 0.4 mg/ml soaked sponge applied to sclera (for up to 2 min) after flap is made during trabeculectomy surgery.
  Mytomycin C 0.4 mg/ml: Mitomycin C 0.4 mg/ml applied with soaked pledget inserted in the sub-tenon's space during glaucoma surgery.
Period: Overall Study
Arm/Group | Treatment 1 (Ranibizumab 0.5mg) | Treatment 2 (Mitomycin C 0.4 mg/ml)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 (Ranibizumab 0.5mg) | Treatment 2 (Mitomycin C 0.4 mg/ml) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Full Range); unit: Years] | 67 [40 to 85] | 68.5 [42 to 90] | 67.75 [40 to 90]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 11 | 8 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Percentage of participants with ocular adverse events and other adverse events as identified by eye examination, physical examination, subject reporting and changes in vital signs one year post-operatively.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment 1 (Ranibizumab 0.5mg) | Treatment 2 (Mitomycin C 0.4 mg/ml)
Number analyzed (Participants) | 12 | 12
percentage of participants | 100 | 16.67

2. Secondary Outcome: Post-Operative Requirement for Glaucoma Medication
Description: Mean number of glaucoma medications used by each participant over the course of one year post-operatively.
Time Frame: 1 day, 2 wks, 1, 3, 6 and 12 months
Measure: Mean (95% Confidence Interval); unit: number of glaucoma medications used
Groups:
- B: Mitomycin C 0.4 mg/ml Sponge: Mitomycin C 0.4 mg/ml soaked sponge applied to sclera (for up to 2 min) after flap is made during trabeculectomy surgery. This is the typical method used as an antifibrotic agent.
  Mitomycin C 0.4 mg/ml: Mitomycin C 0.4 mg/ml applied with soaked pledget inserted in the sub-tenon's space during glaucoma surgery.
Arm/Group | A: Ranibizumab 0.5mg (0.05mL) Injection | B: Mitomycin C 0.4 mg/ml Sponge
Number analyzed (Participants) | 12 | 12
number of glaucoma medications used
  1 Day | 0.01 [0.0 to 0.20] | 0.0 [0.0 to 0.05]
  2 wks | 0.0 [0.0 to 0.11] | 0.01 [0.0 to 0.10]
  1 month | 0.13 [0.0 to 0.46] | 0.01 [0.0 to 0.10]
  3 months | 0.66 [0.22 to 1.33] | 0.08 [0.0 to 0.26]
  6 months | 0.34 [0.05 to 0.89] | 0.06 [0.0 to 0.24]
  12 months | 0.15 [0.0 to 0.57] | 0.06 [0.0 to 0.22]

ADVERSE EVENTS:
Description: At each of the six post-operative follow-up visits, patients were assessed for visual acuity, intraocular pressure, anterior chamber depth, optic disc swelling, choroidal detachment, choroidal folds, macular/retinal folds, and needing of the bleb.
Arm/Group | Treatment 1 (Ranibizumab 0.5mg) | Treatment 2 (Mitomycin C 0.4 mg/ml)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (Ranibizumab 0.5mg) (N=12) | Treatment 2 (Mitomycin C 0.4 mg/ml) (N=12)
optic nerve swelling (Eye disorders) | 2 | 0
choroidal detachment (Eye disorders) | 3 | 1
choroidal folds (Eye disorders) | 1 | 0
macular/retinal folds (Eye disorders) | 1 | 0
needling of the bleb (Eye disorders) | 5 | 1

LIMITATIONS AND CAVEATS:
Small sample size. Different surgical techniques among multiple surgeons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No